CLINICAL TRIAL: NCT02975869
Title: Randomized Trial of a Collaborative Palliative and Oncology Care Model for Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: A Collaborative Palliative and Oncology Care Model for Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-439
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Leukemia Care (Active Comparator): Standard Leukemia care
  Interventions: Other: Standard Leukemia Care
- Collaborative Palliative and Oncology Care (Experimental): Collaborative care from Palliative Care and Leukemia will be given
  Interventions: Other: Palliative Care

INTERVENTIONS:
Other: Standard Leukemia Care
  Arms: Standard Leukemia Care
Other: Palliative Care
  Arms: Collaborative Palliative and Oncology Care

SUMMARY:
This research study is evaluating the impact a collaborative palliative care and oncology team will have on the quality of life, symptoms, mood, and end of life outcomes of patients with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). Palliative care is a medical specialty focused on lessening (or "palliating") symptoms and assisting in coping with serious illness.

DETAILED DESCRIPTION:
The main purpose of this study is to compare two types of care - standard leukemia oncology care and standard leukemia oncology care with collaborative involvement of palliative care clinicians to see which is better for improving the experience of patients and families with AML and MDS undergoing treatment.

The investigators aim to find out whether introducing patients and families undergoing AML and MDS treatment to the palliative care team that specializes in symptom management can improve the physical and psychological symptoms that patients and families experience during their hospitalizations for their leukemia care as well as enhance the quality of patients' end of life care.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with high-risk AML, defined as:
* Newly diagnosed patients with AML ≥ 60 years of age
* Newly diagnosed AML with antecedent hematologic disorder
* Newly diagnosed therapy-related AML
* Relapsed AML
* Primary refractory AML

Exclusion Criteria:

* Patients already receiving palliative care
* Major psychiatric illness or comorbid conditions prohibiting compliance with study procedures.
* A diagnosis of acute promyelocytic leukemia (APML)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Patients' quality of life as measured by (FACT-Leukemia) Score at Week-2 Between Study Arms | 2 weeks
  We will compare patients' FACT-Leukemia scores at week-2 adjusting for baseline scores. FACT-Leukemia ranges from 0-176 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Compare patient quality of life longitudinally using FACT-Leukemia Scores longitudinally Between Study Arms. | up to 6 months
  We will compare FACT-leukemia scores longitudinally between study arm. FACT-Leukemia ranges from 0-176 with higher scores indicating better quality of life.
Compare psychological distress (as measured by the Hospital Anxiety and Depression Scale) between Study Arms | up to 6 months
  We will compare patients' psychological distress using the HADS between study arms at week-2 and longitudinally between study arms. The HADS consistent of two subscales assessing anxiety and depression symptoms with scores ranging from 0-21 with higher scores indicating worse psychological distress.
Compare Symptom Burden (as per ESAS) Between Study Arms. | up to 6 months
  We will compare patients' symptom burden using the Edmonton Symptom Assessment Scale (ESAS) between the two arms at week-2 and longitudinally. The ESAS ranges from 0-100 with higher scores indicating worse symptom burden.
Compare Patient-Reported PTSD (as per PTSD-Checklist) between study arms | up to 6 months
  We will compare PTSD symptoms as measured by the PTSD-Checklist (PCL) between the two groups at week-2 and longitudinally. PCL scores range from 17-85 with higher scores indicating worse PTSD symptoms
Compare Patient-Report Of Discussion EOL Care Preferences Between Study Arms | up to 6 months
  We will compare patient-reported discussing their EOL care preferences between the two groups
Compare Rates Of Chemotherapy Administration Within 30 Days Of Death Between The Two Study Arms | up to 6 months
  to compare rates of chemotherapy administration near the end of life between the two arms
Compare Rates Of Hospitalizations Within 7 Days Of Death Between The Study Arms | up to 6 months
  to compare rates of hospitalizations within the last week of life between the study arms
Compare Rates Of Hospice Utilization And Length-Of-Stay In Hospice At The EOL Between The Study Arms. | up to 6 months
  to compare rates of hospice utilization and length-of-stay in hospice at the end of life between the two study arms

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts general Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen-Battaglia M, Sohn MB, Consagra W, Wang Y, Zhang Z, LoCastro M, Davis J, Buettner K, Mortaz S, El-Jawahri AR, Loh KP. Trajectories of physical well-being among adults with acute myeloid leukemia. Blood Adv. 2024 Jun 11;8(11):2612-2621. doi: 10.1182/bloodadvances.2023011804. PMID 38429079
- [Derived] El-Jawahri A, LeBlanc TW, Kavanaugh A, Webb JA, Jackson VA, Campbell TC, O'Connor N, Luger SM, Gafford E, Gustin J, Bhatnagar B, Walker AR, Fathi AT, Brunner AM, Hobbs GS, Nicholson S, Davis D, Addis H, Vaughn D, Horick N, Greer JA, Temel JS. Effectiveness of Integrated Palliative and Oncology Care for Patients With Acute Myeloid Leukemia: A Randomized Clinical Trial. JAMA Oncol. 2021 Feb 1;7(2):238-245. doi: 10.1001/jamaoncol.2020.6343. PMID 33331857